CLINICAL TRIAL: NCT01555645
Title: How Can Health Care Help Female Breastcancer Patients Reduce Their Stress Symptoms? A Randomized Intervention Study With Stepped-care
Brief Title: Stress Management in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K2010-70X-21412-01-3; CAN 2009/25 (Other Grant/Funding Number: the Swedish Cancer Society); CAN 2011/08 (Other Grant/Funding Number: the Swedish Cancer Society)
Record Dates: First submitted 2012-02-28; First posted 2012-03-15 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer; Stress
Keywords: Breast cancer; Stress management; Stepped care; Randomized
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stress management Individual format (Experimental): The methods and techniques will be the same as those used in the group intervention. The first session will be used for a detailed assessment of the individual's psychosocial problems, as used in earlier studies. The sessions will last 45 - 60 minutes. The number of sessions will depend on the individual patient's problems and the joint assessment made by the patient and nurse together. The total number of sessions will be at least 4, with a maximum of 8. The contents of the sessions are Session 1: Assessment, Session 2: Analysis of diary (self-registration) and suggestions for problem management, Session 3: Evaluation of problem management skills Session 4: Follow-up and conclusion of the intervention. When necessary Sessions 5 -8 will address specific obstacles and continued practice.
  Interventions: Behavioral: Stress management, in two steps
- Stress management Group format (Experimental): Participants will meet for 2 hours every week for a total of 20 hours. In the intervals between the group meetings patients will be asked to do homework. Homework entails practicing problem-solving techniques, keeping a diary, practicing relaxation or physical activities. Each group meeting has a specific subject, i.e. What is stress and stress behaviors, Stress related symptoms, How to manage anger and negative thoughts, Self-registrations and behavioral changes, Future perspectives, Cancer, stress and relations, Expectations and demands, Body, pleasure and sexuality.
  Interventions: Behavioral: Stress management, in two steps

INTERVENTIONS:
Behavioral: Stress management, in two steps — All patients start at the first step of the intervention program with a two hours psychoeducation in stress management. Patients, who don't report a decrease in stress related symptoms, after the first step will be offered an intensive stress management, either in individual or group format. Components included in the intervention concern 1) basic knowledge about cancer, treatment, healthy living and stress reactions, 2) self-awareness with help of diary for thoughts, feelings and behavior 3) instruction in various techniques on how to express negative feelings, how to communicate with others more effectively, how to change behaviors related to stress 4) training these techniques in real-life situations 5) cognitive restructuring 6) spirituality, derived from cognitive behavior therapy.

SUMMARY:
The purpose of this study within Caring sciences is to identify women with breast cancer who have stress symptoms and to offer these women appropriate care to reduce stress and increase well-being. This will be achieved by

1. Studying the prevalence of stress related symptoms in female patients with breast cancer
2. Testing the use of two short screening instruments to identify women at risk for developing long-standing stress symptoms
3. Studying the level and intensity of stress management interventions required to achieve increased well-being, using a stepped-care approach.
4. Studying the effects of interventions based on cognitive behavior therapy, delivered individually or in a group format.

The hypothesis is that half of the individuals assigned to a low intensity intervention will be significantly improved after treatment. For individuals who continue to have symptoms after low intensity treatment it is hypothesized that continued treatment in a group setting with high intensity interventions will be more cost-effective. In addition the assumption is that reduction of stress symptoms in women with breast cancer will lead to a reduction in socio-economic costs.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18
* a recent diagnosis of breast cancer
* scheduled for adjuvant treatment in Falun, Gävle or Uppsala (Sweden)

Exclusion Criteria:

* ongoing psychiatric condition
* language deficiencies in Swedish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2009-05; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Psychosocial aspect | Changes in psychosocial aspects from baseline to 12 months post diagnosis
  Intrusion, Avoidance, Anxiety, Depression, Quality of life, Fatigue, Daily stress

SECONDARY OUTCOMES:
Cost-Utility Analysis | 12 month
Patient satisfaction | 3 month, after intensive intervention and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Karin Nordin, Prof, Principal Investigator — Uppsala University
Locations (3):
- Sweden (3):
  - Falun
  - Gävle
  - Uppsala

REFERENCES:
- [Derived] Hellerstedt-Borjesson S, Nordin K, Fjallskog ML, Holmstrom IK, Arving C. Women Treated for Breast Cancer Experiences of Chemotherapy-Induced Pain: Memories, Any Present Pain, and Future Reflections. Cancer Nurs. 2016 Nov/Dec;39(6):464-472. doi: 10.1097/NCC.0000000000000322. PMID 26632880
- [Derived] Nordin K, Rissanen R, Ahlgren J, Burell G, Fjallskog ML, Borjesson S, Arving C. Design of the study: how can health care help female breast cancer patients reduce their stress symptoms? A randomized intervention study with stepped-care. BMC Cancer. 2012 May 4;12:167. doi: 10.1186/1471-2407-12-167. PMID 22559200